CLINICAL TRIAL: NCT04680364
Title: Effects of Ballroom Dance on Physical Fitness and Reaction Time in Experienced Older Adults
Brief Title: Effects of Dance on Reaction Time in Experienced Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, prof. Gian Pietro Emerenziani, Professor, University Magna Graecia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N395/2020
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Aging
Keywords: physical activity; partnered dances; cognitive functions; fall prevention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants (Experimental): to analyze the effects of 6-month ballroom dance (3 times/wk) on physical fitness and reaction time in twenty-four experienced older adults
  Interventions: Other: partnered dance

INTERVENTIONS:
Other: partnered dance — Dance classes consisted of different choreographies, which include rhythmic and simple movements typically of ballroom/standard dances (Waltz, Tango, Viennese Waltz).

SUMMARY:
Aim of this study was to investigate the effects of 6-month ballroom dance (3 times/wk) on physical fitness and reaction time in twenty- four experienced older adults. Body composition, handgrip test, standing long jump test, step test, one-legged stance balance test, and reaction time (RT) test were assessed before and after 6 months (T6) of dance practice. RT was re-evaluated after 4 months (T10).

ELIGIBILITY:
Inclusion Criteria:

* dance practice (dance average years = 11 years)

Exclusion Criteria:

* functional inabilities
* cardiovascular diseases
* prosthesis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Reaction time at 6 Months | baseline, 6 months and 10 months
  reaction time was assessed with the subject seating with the arm resting on a table in a comfortable position and then catches the apparatus as quickly as possible after it begins to fall. The fall distance was measured and it was converted into a reaction time (in milliseconds) using the formula for a body falling under the influence of gravity (d 5 1⁄2gt2), where d is distance, g is acceleration due to gravity, and t is time.

CONTACTS AND LOCATIONS:
Locations (1):
- Dance School "Free Dance", Catanzaro, Calabria, Italy

IPD SHARING:
Plan to Share IPD: No
Scientific dataset will be shared on request

REFERENCES:
- [Result] Vaccaro MG, Izzo G, Ilacqua A, Migliaccio S, Baldari C, Guidetti L, Lenzi A, Quattrone A, Aversa A, Emerenziani GP. Characterization of the Effects of a Six-Month Dancing as Approach for Successful Aging. Int J Endocrinol. 2019 Jun 17;2019:2048391. doi: 10.1155/2019/2048391. eCollection 2019. PMID 31316562
- [Result] Kattenstroth JC, Kalisch T, Holt S, Tegenthoff M, Dinse HR. Six months of dance intervention enhances postural, sensorimotor, and cognitive performance in elderly without affecting cardio-respiratory functions. Front Aging Neurosci. 2013 Feb 26;5:5. doi: 10.3389/fnagi.2013.00005. eCollection 2013. PMID 23447455
- [Result] Kattenstroth JC, Kalisch T, Kolankowska I, Dinse HR. Balance, sensorimotor, and cognitive performance in long-year expert senior ballroom dancers. J Aging Res. 2011;2011:176709. doi: 10.4061/2011/176709. Epub 2011 Sep 25. PMID 21961064